CLINICAL TRIAL: NCT00735930
Title: Phase 1 Trial of Flavopiridol in Combination With Lenalidomide in Patients With Relapsed or Refractory B-Cell CLL/SLL
Brief Title: Lenalidomide and Alvocidib in Treating Patients With Relapsed or Refractory B-cell Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00269; NCI-2009-00269 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU-08056; 2008C0033; CDR0000738866; OSU 08056 (Other: Ohio State University Comprehensive Cancer Center); 8046 (Other: CTEP); P30CA016058 (NIH); U01CA076576 (NIH)
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-02

CONDITIONS: Anemia; Chronic Lymphocytic Leukemia; Prolymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Thrombocytopenia
MeSH Terms: conditions — Anemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic; Thrombocytopenia | interventions — alvocidib; Lenalidomide

ARMS (1):
- Treatment (alvocidib, lenalidomide) (Experimental): Patients receive alvocidib IV over 4.5 hours on days 1, 8, and 15 in course 1 followed by a week of rest. Beginning in course 2 and all subsequent courses, patients receive lenalidomide PO QD on days 1-21 and alvocidib IV over 4.5 hours on days 3, 10, and 17. Treatment repeats every 35 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alvocidib Hydrochloride; Drug: Lenalidomide; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Alvocidib Hydrochloride — Given IV
  Other Names: FLAVO; HL-275; HMR 1275
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; IMiD-1
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of lenalidomide when given together with alvocidib in treating patients with relapsed or refractory B-cell chronic lymphocytic leukemia or small lymphocytic lymphoma. Lenalidomide may stop the growth of leukemia or lymphoma by blocking blood flow to the cancer. Alvocidib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving lenalidomide together with alvocidib may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of flavopiridol (alvocidib) in combination with lenalidomide in patients with relapsed or refractory B-cell chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL).

II. To define the specific toxicities and the dose limiting toxicity (DLT) of flavopiridol in combination with lenalidomide in the treatment of patients with relapsed or refractory CLL/SLL.

SECONDARY OBJECTIVES:

I. To assess preliminary efficacy of flavopiridol combined with lenalidomide in patients with relapsed/refractory CLL/SLL to justify future, rigorous phase II studies of the combination in CLL.

II. To determine the pharmacokinetics of flavopiridol and lenalidomide alone and in combination in patients with CLL/SLL.

III. To correlate select pre-treatment prognostic markers, including interphase cytogenetics with minimal residual disease, progression-free survival, response, and toxicity following combination therapy with flavopiridol and lenalidomide.

IV. To determine patient cytokine expression profiles immediately pre-treatment, after flavopiridol dosing, and after combination flavopiridol and lenalidomide therapy to assess the impact of lenalidomide on flavopiridol induced cytokine release (interleukin [IL]-6).

V. To assess if pre-treatment ex vivo and in vivo (day 1 and day 3 of lenalidomide) immune (B-cell, natural killer [NK] cell, and T-cell) activation correlates with response and toxicity of lenalidomide therapy.

VI. To assess the in vivo effect of lenalidomide on flavopiridol on the modulation of selected intracellular pharmacodynamic targets including signal transducer and activator of transcription 3 (acute-phase response factor) (STAT3), myeloid cell leukemia sequence 1 (BCL2-related) (Mcl-1), and other downstream IL-6 targets.

OUTLINE: This is a dose-escalation study of lenalidomide.

Patients receive alvocidib intravenously (IV) over 4.5 hours on days 1, 8, and 15 in course 1 followed by a week of rest. Beginning in course 2 and all subsequent courses, patients receive lenalidomide orally (PO) once daily (QD) on days 1-21 and alvocidib IV over 4.5 hours on days 3, 10, and 17. Treatment repeats every 35 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed B-cell CLL/SLL according to World Health Organization (WHO) criteria, or B-cell prolymphocytic leukemia (B-PLL) arising from CLL with at least one of the following indications for treatment:

  * Progressive disease or marked splenomegaly and/or lymphadenopathy
  * Anemia (hemoglobin < 11 mg/dL) or thrombocytopenia (platelets < 100,000/mm^3)
  * Unexplained weight loss exceeding 10% of body weight over the preceding 6 months
  * National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v 4.0) grade 2 or 3 fatigue
  * Fevers > 100.5 or night sweats for greater than 2 weeks without evidence of infection
  * Progressive lymphocytosis, with an increase exceeding 50% over a 2 month period or a doubling time of less than 6 months
* Must have at least one prior therapy that includes either fludarabine (or equivalent nucleoside analogue) or an alternative regimen if a contra-indication to fludarabine exists (i.e., autoimmune hemolytic anemia); prior therapy with flavopiridol is not permitted; prior lenalidomide is permitted provided that it has been > 6 months since the last lenalidomide dose
* Eastern Cooperative Oncology Group (ECOG) performance status =< (Karnofsky >= 60%)
* White blood cell count =< 150,000/mm^3
* Absolute neutrophil count >= 1,000/mm^3
* Platelets >= 30,000/mm^3
* Total bilirubin =< 1.5 X institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamate pyruvate transaminase (SGPT) =< 2.5 X institutional ULN
* Creatinine =< 1.5 mg/dL OR creatinine clearance >= 60 ml/min
* Recovery to =< grade 1 from all toxicities associated with prior therapy
* Not pregnant or breast-feeding; woman of child bearing potential should have a negative pregnancy test (serum beta-human chorionic gonadotropin [HCG]) within 7-14 days of starting cycle 1 of treatment; woman of child bearing potential should have a negative pregnancy test (serum beta-HCG) within 10-14 days of starting cycle 2, the start of lenalidomide treatment (i.e. days 14-18 of cycle 1), and an additional test within 24 hours of starting cycle 2 treatment
* Patient must agree to use adequate contraception for 4 weeks prior to the start of lenalidomide and up to 28 days following the last dose of lenalidomide to avoid risk of pregnancy

  * Women of child-bearing potential will be required to use two methods of birth control; one "highly effective method" and one "additional effective method" as defined below:

    * Highly effective methods

      * Intrauterine device
      * Hormonal (oral contraceptive, implants)
      * Tubal ligation
      * Partner's vasectomy
      * Abstinence
    * Alternative effective methods

      * Latex condoms
      * Diaphragm
      * Cervical cap
  * Men must agree to use latex condoms
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days and again within 24 hours prior to starting cycle 1 of lenalidomide; further, they must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP, even if they have had a successful vasectomy; all patients must be counseled by a trained counselor every 28 days about pregnancy precautions and risks of fetal exposure
* Patients must agree not to donate blood, semen, sperm/ova during the course of taking lenalidomide and for 28 days after stopping lenalidomide treatment
* Patients must have the ability to understand and the willingness to sign a written informed consent document
* Patients who are glucose-6-phosphate dehydrogenase (G6PD) deficient are not eligible for this study
* Only human immunodeficiency virus (HIV)-positive patients meeting all of the following criteria may be enrolled on this trial:

  * Cluster of differentiation (CD) 4 count > 500/mm^3
  * Not receiving highly active anti-retroviral therapy (HAART) or anti-HIV viral therapy
  * HIV viral load < 10,000 HIV messenger ribonucleic acid (mRNA) copies/mm^3
  * No history of acquired immune deficiency syndrome (AIDS)-defining illness

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated on this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-08; Primary Completion 2013-03 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
MTD of lenalidomide when combined with alvocidib, defined as the maximum dose level with fewer than 2 of 6 patients experiencing dose limiting toxicity (DLT) | Up to day 70
Incidence of DLT in patients treated with alvocidib and lenalidomide graded according to NCI CTCAE version 4.0 | Up to day 70
  Toxicities classified as DLT during course 1 will not be considered DLT for the combination of lenalidomide and flavopiridol, but will result in patient removal from the study.

SECONDARY OUTCOMES:
Pharmacokinetic parameters of alvocidib and lenalidomide alone and in combination in plasma samples | Baseline, day 1 of course 1, and on days 2-3 of course 2
  Samples will be analyzed in batches to assess plasma drug concentrations, the plasma drug concentration-time profile (AUC), volume of distribution (Vss), clearance (CL), and half-life. Standard paired statistical tests, parametric and nonparametric, will be used to compare baseline with treatment values. With data collected serially over time, repeated measures analysis of variance will be used to analyze data.
Plasma IL-6 and selected cytokine levels | Up to 5 years
  Standard paired statistical tests, parametric and nonparametric, will be used to compare baseline with treatment values. With data collected serially over time, repeated measures analysis of variance will be used to analyze data.
B-cell activation as assessed by surface antigen (CD40, CD80, CD86, HLA-DR, and CD95) expression | Up to 5 years
  Standard paired statistical tests, parametric and nonparametric, will be used to compare baseline with treatment values. With data collected serially over time, repeated measures analysis of variance will be used to analyze data.
Intracellular pharmacodynamic targets including STAT3, Mcl-1, and nuclear factor kappa-light-chain-enhancer of activated B cells (NF-kB) | Up to 5 years
  Standard paired statistical tests, parametric and nonparametric, will be used to compare baseline with treatment values. With data collected serially over time, repeated measures analysis of variance will be used to analyze data.
Response assessed by National Cancer Institute-Sponsored Working Group guidelines | Up to 5 years
  Standard paired statistical tests, parametric and nonparametric, will be used to compare baseline with treatment values. With data collected serially over time, repeated measures analysis of variance will be used to analyze data.
Progression-free survival (PFS) | Time from start of treatment to time of progression, assessed up to 5 years
  Standard paired statistical tests, parametric and nonparametric, will be used to compare baseline with treatment values. With data collected serially over time, repeated measures analysis of variance will be used to analyze data.
Toxicity graded according to NCI CTCAE version 4.0 | Up to 5 years
  Standard paired statistical tests, parametric and nonparametric, will be used to compare baseline with treatment values. With data collected serially over time, repeated measures analysis of variance will be used to analyze data.
Presence of minimal residual disease | Up to 5 years
  Standard paired statistical tests, parametric and nonparametric, will be used to compare baseline with treatment values. With data collected serially over time, repeated measures analysis of variance will be used to analyze data.

CONTACTS AND LOCATIONS:
Overall Officials: Kristie Blum, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States